CLINICAL TRIAL: NCT00039910
Title: Safety and Efficacy of (PN-152,243)/PN-196,444 in the Prevention of Thrombocytopenia in Recurrent or Refractory Non-Burkitt's, Non-Hodgkin's Lymphoma (NHL) or Hodgkin's Disease Receiving DHAP (Dexamethasone, High-Dose Cytarabine and Cisplatin) Chemotherapy
Brief Title: Safety and Efficacy of (PN-152,243)/PN-196,444 in the Prevention of Thrombocytopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444-ONC-0003-0019
Record Dates: First submitted 2002-06-14; First posted 2002-06-17 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2006-09

CONDITIONS: Non-Hodgkin Lymphoma; Hodgkin Disease; Thrombocytopenia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Thrombocytopenia

INTERVENTIONS:
Drug: (PN-152,243)/ PN-196,444

SUMMARY:
Intensive chemotherapy is associated with significant thrombocytopenia, often requiring platelet transfusion to maintain platelet counts. This investigational drug has been demonstrated to increase platelet counts. This study will test the safety and efficacy of the investigational drug in the prevention of thrombocytopenia in patients with recurrent or refractory intermediate-grade or high-grade non-Burkitt's, non-Hodgkin's lymphoma (NHL), or Hodgkin's disease receiving DHAP (Dexamethasone, high-dose Cytarabine, and Cisplatin) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or refractory intermediate-grade or high-grade non-Burkitt's, non-Hodgkin's lymphoma (NHL) or Hodgkin's disease and be scheduled for a minimum of 2 cycles of DHAP (Dexamethasone, high-dose Cytarabine and Cisplatin) chemotherapy

Exclusion Criteria:

* Patients must not have active bleeding (exclusions do apply) or history of platelet disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2000-07; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of primary prophylaxis with intravenous rhTPO versus placebo in reducing the cumulative proportion of patients who experience severe chemotherapy-induced thrombocytopenia.

SECONDARY OUTCOMES:
Identify the effect of rhTPO on the number of platelet transfusions
Evaluate the severity and duration of thrombocytopenia and neutropenia associated with rhTPO prophylaxis
Quantify the effect of rhTPO on the occurrence of any bleeding events associated with thrombocytopenia
Assess the likelihood that patients were to have adequate hematologic recovery to allow on-time chemotherapy administration in the subsequent cycles
Assess the safety of multiple IV doses of rhTPO
Determine the occurrence and clinical implications of any anti-TPO antibodies
Assess the antitumor activity of DHAP chemotherapy
Evaluate the impact of rhTPO prophylaxis on health economics/cost effectiveness
Evaluate the impact of rhTPO prophylaxis on patient quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (21):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Tamarac, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Saint Joseph, Michigan
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Coos Bay, Oregon
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Abingdon, Virginia
  - Pfizer Investigational Site, Lebanon, Virginia
  - Pfizer Investigational Site, Marion, Virginia
- Pfizer Investigational Site, East Melbourne, Victoria, Australia
- France (2):
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Tours
- Pfizer Investigational Site, Thessaloniki, Macedonia, Greece
- Pfizer Investigational Site, Shatin, New Territories, Hong Kong
- Poland (2):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Warsaw
- Pfizer Investigational Site, Moscow, Russia
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=444-ONC-0003-0019&StudyName=Safety+and+Efficacy+of+%28PN%2D152%2C243%29%2FPN%2D196%2C444+in+the+Prevention+of+Thrombocytopenia